CLINICAL TRIAL: NCT04907747
Title: Efficacy and Safety of Furazolidone-based Quadruple Therapy With Vonoprazan as First-line Treatment for Helicobacter Pylori Eradication: A Prospective Randomized Trial
Brief Title: Efficacy and Safety of Vonoprazan as First-line Treatment for Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0446
Record Dates: First submitted 2021-05-24; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; vonoprazan
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole; Amoxicillin; Furazolidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Vonoprazan taken with bismuth, amoxicillin, furazolidone for 10 days (Experimental): Vonoprazan 20mg qd, Colloidal bismuth pectin 200mg bid, Amoxicillin 1.0g bid, Furazolidone 0.1g bid for 10days
  Interventions: Drug: Vonoprazan; Drug: Colloidal bismuth pectin; Drug: Amoxicillin; Drug: Furazolidone
- Group B: Vonoprazan taken with bismuth, amoxicillin, furazolidone for 14 days (Experimental): Vonoprazan 20mg qd, Colloidal bismuth pectin 200mg bid, Amoxicillin 1.0g bid, Furazolidone 0.1g bid for 14days
  Interventions: Drug: Vonoprazan; Drug: Colloidal bismuth pectin; Drug: Amoxicillin; Drug: Furazolidone
- Group C: Esomeprazole taken with bismuth, amoxicillin, furazolidone for 14 days (Active Comparator): Esomeprazole 20 mg bid, Colloidal bismuth pectin 200mg bid, Amoxicillin 1.0g bid, Furazolidone 0.1g bid for 14days
  Interventions: Drug: Esomeprazole; Drug: Colloidal bismuth pectin; Drug: Amoxicillin; Drug: Furazolidone

INTERVENTIONS:
Drug: Vonoprazan — Potassium-competitive acid blocker
  Arms: Group A: Vonoprazan taken with bismuth, amoxicillin, furazolidone for 10 days; Group B: Vonoprazan taken with bismuth, amoxicillin, furazolidone for 14 days
Drug: Esomeprazole — Proton pump inhibitor
  Arms: Group C: Esomeprazole taken with bismuth, amoxicillin, furazolidone for 14 days
Drug: Colloidal bismuth pectin — Gastric mucosal protective drug with anti-H. pylori effect
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: Furazolidone — Antibiotic for H. pylori eradication

SUMMARY:
This study aims to evaluate the efficacy of vonoprazan compared with esomeprazole as first-line treatment for Helicobacter Pylori(Hp) eradication, as well as the safety and economic benefits.

DETAILED DESCRIPTION:
Vonoprazan, a novel potassium-competitive acid blocker, is proved to be superior to proton pump inhibitor in gastric acid-related diseases such as reflux esophagitis, as the increase of intragastric pH maintains for a longer period. Vonoprazan, therefore, is a promising candidate in helicobacter pylori eradication as the antibiotic resistance is rising.

This study will enroll 234 patients, and randomly assigned by computer to one of the three treatment groups.

Group A: Vonoprazan taken with bismuth, amoxicillin, furazolidone for 10 days Group B: Vonoprazan taken with bismuth, amoxicillin, furazolidone for 14 days Group C: Esomeprazole taken with bismuth, amoxicillin, furazolidone for 14 days Participants will visit the clinic for a follow-up assessment 6-8 weeks after the course of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Helicobacter pylori-positive participants determined by ¹³C-urea breath test, ¹⁴C-urea breath test, HE stain or bacterium culture
2. With no historical treatment for helicobacter pylori infection.

Exclusion Criteria:

1. Administration of antibiotics, bismuth in 4 weeks prior to inclusion or antacids including H2 receptor antagonist, proton pump inhibitor and potassium-competitive acid blocker in 2 weeks prior to inclusion
2. Active peptic ulcer with complications such as hemorrhage, perforation, obstruction, cancerization, etc.
3. With previous esophageal or gastric surgery
4. With severe systemic diseases, major organ like heart, lung, brain diseases, liver or kidney insufficiency, malignant tumor or other diseases
5. Allergy to any of the study drugs
6. Pregnancy or in lactation
7. Participated in other research within 3 months，cannot express his/her own ideas correctly or cannot cooperate with the researcher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-05-18 (Estimated); Primary Completion 2022-04-13 (Estimated); Study Completion 2022-04-13 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori Eradication Rate | Six to eight weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by ¹³C-urea breath test six to eight weeks after completion of the medication.

SECONDARY OUTCOMES:
Rate of Adverse Drug Reaction(ADR) | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types (with mnemonics): dose-related (Augmented), non-dose-related (Bizarre), dose-related and time-related (Chronic), time-related (Delayed), withdrawal (End of use), and failure of therapy (Failure).
Compliance Rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Lu L, Wang Y, Ye J, Han Y, Lou G, Li Y, Yan H, Du Q. Quadruple therapy with vonoprazan 20 mg daily as a first-line treatment for Helicobacter pylori infection: A single-center, open-label, noninferiority, randomized controlled trial. Helicobacter. 2023 Feb;28(1):e12940. doi: 10.1111/hel.12940. Epub 2022 Dec 1. PMID 36458325